CLINICAL TRIAL: NCT02744157
Title: Long Term Effects on Lifestyle Habits and Quality of Life in Individuals With Increased Cardiometabolic Risk Participating in a Structured Lifestyle Intervention Program
Brief Title: Long Term Effects of a Structured Lifestyle Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Mai-Lis Hellenius, Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015/494-31/2
Record Dates: First submitted 2016-03-03; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Lifestyle; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- structured lifestyle program (Other): The program consisted of an individual visit to a nurse for a health check-up and lifestyle counseling at baseline, six month and one year. The program also consisted of five group educations which included lectures on nicotine, alcohol, physical inactivity, eating habits, stress, sleeping habits and behavior changes
  Interventions: Behavioral: Longterm effects after a structured lifestyle program

INTERVENTIONS:
Behavioral: Longterm effects after a structured lifestyle program — present study was to describe a structured intervention to reduce cardiovascular risk in a clinical setting and to study the effects of the program on lifestyle habits and quality of life in individuals at risk after six months and one year.

SUMMARY:
The aim of the present study was to describe a structured intervention to reduce cardiovascular risk in a clinical setting and to study the effects of the program on lifestyle habits and quality of life in individuals at risk after six months and one year.

ELIGIBILITY:
Inclusion criteria:

(three risk factors )

* cardiovascular disease
* physical inactivity
* smoking
* risk consumption of alcohol
* unhealthy food habits
* stress
* overweight or abdominal obesity
* high lipids (cholesterol, LDL)
* high blood pressure
* diabetes/insulin resistance.

Exclusion criteria:

* Not understand Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk | change from baseline in waist circumference after one year
  change from baseline in waist circumference after one year

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Lis Hellenius, Professor, Principal Investigator — Karolinska Institutet, Department of medicine and Karolinska University Hospital,Department of Cardiology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lidin M, Hellenius ML, Rydell-Karlsson M, Ekblom-Bak E. Long-term effects on cardiovascular risk of a structured multidisciplinary lifestyle program in clinical practice. BMC Cardiovasc Disord. 2018 Apr 2;18(1):59. doi: 10.1186/s12872-018-0792-6. PMID 29609555